CLINICAL TRIAL: NCT03020537
Title: U19 Influenza Immunity: Protective Mechanisms Against a Pandemic Respiratory Virus. Project 1: B-cell Immunity to Influenza. Technical Development Project 1: Measuring the Immunome: Genomic Approaches to B-cell Repertoire- Year 5, 2013
Brief Title: B-cell Immunity to Influenza (SLVP017)- Year 5, 2013
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Study Principal Investigator, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SU-17218-2013; 2U19AI057229-06 (NIH)
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Influenza
Keywords: Trivalent inactivated influenza vaccine; Young children; Young adults
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: 1-2 years old (Other): Group A: 1-2 years old, seasonal influenza vaccine-naive. Given intramuscular,inactivated influenza vaccine-trivalent (IM IIV3) - Fluzone (pediatric formulation).
  Interventions: Biological: Fluzone
- Group B: 18-30 years old (Other): Group B: 18-30 years old, who did not receive the 20l2-2013 seasonal influenza vaccine. Given intramuscular,inactivated influenza vaccine-trivalent (IM IIV3) - Fluzone.
  Interventions: Biological: Fluzone

INTERVENTIONS:
Biological: Fluzone — Fluzone (Influenza Virus Vaccine) Suspension for Intramuscular Injection 2013-2014 Formula.

SUMMARY:
In this exploratory study, investigators will be looking at immune response differences between age groups and between the two different vaccines given to identical twins and vaccine-naive young adults.

DETAILED DESCRIPTION:
This is a study of healthy children and adults who will be given standard seasonal influenza vaccination (IIV3). There are no exclusions for gender, ethnicity or race. Following review and confirmation of written informed consent, volunteers will be enrolled into the study.

The 1-2 year-old child volunteers enrolled in Group A cannot have been previously immunized with an influenza vaccine. They will receive two single doses of the 2013-2014 pediatric formulation of seasonal trivalent inactivated influenza vaccine (IIV3), at least 28 days apart, given by intramuscular (IM) injection. The child volunteers will complete 4 clinic visits with 3 blood sample collections. Study visits will be on Day 0 (first immunization), Day 28-32 (second immunization), Day 6-8 post-Dose 2, and Day 28+4 post-Dose 2. The baseline blood sample will be drawn prior to immunization at Day 0, followed by two additional blood samples at Day 6-8 post-Dose 2, and Day 28+4 post-Dose 2. There will not be a blood sample collected at Day 28-32.

The 18-30 year-old young adults in Group B cannot have been immunized with the 2012-2013 seasonal influenza vaccine. Participants in Group B will receive a single dose of the 2013-2014 IIV3 by IM injection. Young adult volunteers will complete 3 clinic visits with 3 blood sample collections on Day 0, Day 6-8, and Day 28+4. The baseline blood sample will be drawn prior to immunization at Day 0.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, ambulatory children 1-2 years of age or 18-30 year-old young adults.
2. Willing to complete the informed consent process.
3. Availability for follow-up for the planned duration of the study (after last study immunization, approximately 8 weeks for Group A and 4 weeks for Group B).
4. Acceptable medical history by medical history and vital signs.

Exclusion Criteria:

1. Group A: Prior vaccination with a seasonal flu vaccine (IIV). Group B: Prior vaccination with the 2012-2013 seasonal flu vaccine (IIV or LAIV).
2. Prior off-study vaccination with the current 2013-2014 seasonal IIV or LAIV
3. Allergy to egg or egg products, or to vaccine components.
4. Life-threatening reactions to previous influenza vaccinations
5. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
6. History of immunodeficiency (including HIV infection)
7. Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease, or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
8. Chronic Hepatitis B or C.
9. Recent or current use of immunosuppressive medication, including systemic glucocorticoids (corticosteroid nasal sprays and topical steroids are permissible; use of inhaled steroids, or oral steroids (<20mg prednisone-equivalent/day), may be acceptable after review by the investigator.
10. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
11. Autoimmune disease (including rheumatoid arthritis) treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
12. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
13. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except up to 325 mg. per day), Plavix, or Aggrenox must be reviewed by investigator to determine if this would affect the volunteer's safety.
14. Receipt of blood or blood products within the past 6 months
15. Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
16. Inactivated vaccine within 14 days prior to study vaccination (inform study staff of any non-study vaccinations received during study period)
17. Live, attenuated vaccine within 30 days prior to first study vaccination, or planned immunization with a live, attenuated vaccine before completion of study visits (inform study staff of any non-study vaccinations received during study period).
18. Need for allergy immunizations (that cannot be rescheduled if necessary) during the study period
19. History of Guillain-Barre Syndrome
20. Pregnant or lactating woman
21. Use of investigational agents within 30 days prior to enrollment or planned use of investigational agents prior to completion of study visits
22. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment
23. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Dekker, MD, Principal Investigator — Stanford University; Harry Greenberg, MD, Principal Investigator — Stanford University; Stephen Quake, PhD, Principal Investigator — Stanford University; Xiaosong He, PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le Gars M, Kay AW, Bayless NL, Aziz N, Dekker CL, Swan GE, Davis MM, Blish CA. Increased Proinflammatory Responses of Monocytes and Plasmacytoid Dendritic Cells to Influenza A Virus Infection During Pregnancy. J Infect Dis. 2016 Dec 1;214(11):1666-1671. doi: 10.1093/infdis/jiw448. Epub 2016 Sep 21. PMID 27655870

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: 1 - 2 Years Old: Group A: 1-2 years old, seasonal influenza vaccine-naive. Given intramuscular,inactivated influenza vaccine-trivalent (IM IIV3) - Fluzone (pediatric formulation).
  Fluzone: Fluzone (Influenza Virus Vaccine) Suspension for Intramuscular Injection 2013-2014 Formula.
Period: Overall Study
Arm/Group | Group A: 1 - 2 Years Old | Group B: 18-30 Years Old
Started | 1 | 7
Completed | 1 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: 1 - 2 Years Old | Group B: 18-30 Years Old | Total
Number analyzed (Participants) | 1 | 7 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.128 (0) | 27.29 (4.066) | 24.025 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 1 | 5 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 5 | 5
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 7 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received Influenza Vaccine
Time Frame: Day 0 to 28
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 1 - 2 Years Old | Group B: 18-30 Years Old
Number analyzed (Participants) | 1 | 7
Participants | 1 | 7

2. Secondary Outcome: Number of Participants With Related Adverse Events
Time Frame: Day 0 to 28 post-immunization
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 1 - 2 Years Old | Group B: 18-30 Years Old
Number analyzed (Participants) | 1 | 7
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Day 0 to 28 of study participation
Description: Clinical Assessment performed at each visit
Arm/Group | Group A: 1 - 2 Years Old | Group B: 18-30 Years Old
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/7
Other Adverse Events (participants affected / at risk) | 1/1 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: 1 - 2 Years Old (N=1) | Group B: 18-30 Years Old (N=7)
Erythema at vaccination site 0.5 cm (General disorders) | 1 (1) | 1 (1) — Erythema at vaccination site after dose 2
Mild Pruritus at Vaccination site Right Deltoid (General disorders) | 0 (0) | 1 (1) — Mild Pruritus at Vaccination site Right Deltoid

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No